CLINICAL TRIAL: NCT06524180
Title: Can TElemedicine System Replace Doctor Consultations to Achieve Non-inferior Blood Pressure in Patients With Controlled Hypertension (TEACH)? a Randomised Controlled Trial and Cost-minimization Analysis
Brief Title: Can TElemedicine System Replace Doctor Consultations to Achieve Non-inferior Blood Pressure in Patients With Controlled Hypertension
Acronym: TEACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical associate professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.525
Record Dates: First submitted 2024-07-16; First posted 2024-07-29 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
Keywords: blood pressure; telemedicine; home blood pressure measurement
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): Patients will be (i) given a validated HBPM device (ORMON HEM-7120) with appropriate cuff size, (ii) taught the HBPM technique, and (iii) taught to record HBPM readings using the HealthCap mobile app on their smartphones.
  Participants randomized to intervention will be reminded to take dual BP readings in the morning and evening for 1-2 weeks before the index consultation. These BP readings will be automatically sent to a computer at the clinic. When the HBPM mean is optimal (i.e., <135/85 mmHg or <130/80 mmHg [for patients with cardiovascular diseases, renal diseases, and DM]), other parameters will be checked using an online questionnaire. If no complaints are identified, the patient will have automatic drug refill and the physician appointment will be deferred for 16-18 weeks.
  Interventions: Device: Telemedicine
- Usual care (Active Comparator): Participants will continue receiving routine care, including anti-HT drug prescriptions, from their regular clinicians. In HK, patients with well-controlled HT are routinely seen every 16-18 weeks. Participants will also be given the same HBPM devices and taught the techniques. This is necessary because HBPM is a secondary outcome. According to the HK guidelines, all patients with HT are advised to regularly monitor their home BP, which can be considered as usual care.14 However, the patients will not be taught any BP measurement algorithm (such as that used in the telemedicine group). They will also be asked not to download or use any new HT mobile apps during the study period. In HK, all citizens have unlimited access to GOPCs and emergency departments for health problems. All participants are advised to seek medical help if BP becomes dangerously and persistently high (i.e. SBP ≥180 or DBP ≥110mmHg) or in case of any suspected medical emergencies.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Telemedicine — a mobile app and telemedicine platform to confirm good blood pressure control and may save doctor face-to-face consultation
  Arms: Telemedicine
Other: Usual care — Participants will be followed up as usual by face-to-face consultation with the doctors
  Arms: Usual care

SUMMARY:
The goal of this clinical trial is to evaluate whether patients assigned to the telemedicine (HealthCap) group demonstrate non-inferior blood pressure (BP) control compared to patients in the usual care group at 12 months. The main question it aims to answer is:

* Do participants in telemedicine group have non-inferior daytime ambulatory blood pressure readings at 12-month, compared to usual care group?
* Do participants in telemedicine group have better HT treatment, higher self-efficacy, reduced number of visits to primary care clinics and similar health care utilisation other than GOPCs, compared to usual care group?

Participant in telemedicine group will:

* Receive reminders to measure 7-day home blood pressure before their index consultation.
* Get their drug refilled automatically as well as have consultations deferred 16-18 weeks later, if their blood pressure is under optimal control.
* Have consultations as scheduled, if their BP is suboptimal or any of the safety questions screen positive.

Participants in control group will:

* Have consultation with physicians every 16-18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* (i) having a diagnosis of essential HT;
* (ii) on anti-HT medications;
* (iii) well-controlled HT on out-of-office BP measurements, including HBPM or ambulatory blood pressure measurements (ABPM) (measurement algorithm and details under methods). ABPM or HBPM are preferred to office BP due to their superior reproducibility and predictivity to cardiovascular outcomes. Furthermore, office BP misclassifies 30-40% of patients as having suboptimal BP control due to white-coat effect. From our pilot study, some patients with optimal BP are reluctant to undergo ABPM before recruitment into the RCT, and HBPM is more acceptable to these patients and is therefore included. According to local and international guidelines, optimal out-of-office daytime BP should be <135/85 mmHg for patients without comorbidities and <130/85 mmHg for patients with comorbidities that increase cardiovascular risk (i.e. stroke, ischaemic heart diseases, heart failure, diabetes mellitus (DM), and chronic kidney diseases) respectively;
* (iv) can read basic Chinese (language used in the HealthCap);
* (v) have used any mobile app (not HT-related) in the previous 1 year; and
* (vii) aged between 18-80.

Exclusion Criteria:

* (i) cannot provide informed consent;
* (ii) unwillingness to conduct HBPM or repeated ABPM;
* (iii) relative contraindications to ABPM (i.e., diagnosed atrial fibrillation, nighttime workers, occupational drivers, or patients with bleeding tendencies);
* (iv) have severe mental illnesses that impair their ability to use HealthCap, including those diagnosed with schizophrenia, dementia, or as being actively suicidal;
* (v) a diagnosis of other acute or chronic diseases that need regular physical assessments and/or medication changes (e.g., suboptimally controlled DM [e.g., glycosylated haemoglobin (HbA1c)≥7%], depression requiring medications, active cancer); and (vi) predicted lifespan of <1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
daytime systolic blood pressure | from the enrollment at 12-months
  WatchBP O3 (Microlife AG, Switerzland) has been validated by multiple HT societies (www.stridebp.org) and will be used in the current RCT. BP will be measured every 30 min for ≥24 h, and patients' sleep diary will define the sleep duration. The readings will be considered valid if there are >70% of valid readings overall, >20 valid awake, and >7 valid asleep BP readings in 24-h intervals.

SECONDARY OUTCOMES:
Ambulatory blood pressure readings | from enrollment at 6-month
  This will include ABPM parameters (24-h/daytime/nighttime SBP and DBP)
Ambulatory blood pressure readings | from enrollment at 12-month
  ABPM parameters other than daytime SBP at 12-month (24-h/nighttime SBP/DBP and daytime DBP)
Treatment adherence | from enrollment at 6-month and 12-month
  This will be measured by the Treatment Adherence Questionnaire for patients with HT, which is validated in Chinese, and contains measurements of adherence to medications, diet, stimulation, weight control, exercise, and stress reduction.
Self-efficacy | from enrollment at 6 month and 12 month
  This will be measured using the validated 5-item self-efficacy scale specific to HT, which was found to have good internal validity (Cronbach's alpha = 0.81) with a mean score of at least 9 (out of 10), signifying good self-efficacy.
Satisfaction with HealthCap | from enrollment at 12 month
  all participants in the intervention group will be asked to rank their satisfaction with HealthCap and with the automatic drug refill process on a scale from 0 (completely dissatisfied) to 10 (completely satisfied) at 12-m
Acceptability | from enrollment at 12-month
  to assess the acceptability of the HealthCap system, around 30 patients with high (highest quartile score) and low (lowest quartile score) satisfaction will be invited to patients' interview till data saturation. Similarly, participating physicians (likely total number <30) will be interviewed, till data saturation if possible.
Health-related quality of life | from enrollment at 6-month and 12-month
  Their health-related quality of life will be assessed by the validated EQ5D-5L (needed for cost-effectiveness analysis if HealthCap is found superior than usual care).
serum creatinine | from enrollment at 12 month
  Serum creatinine will be collected to check kidney function
Body weight | from enrollment at 12 month
  Body weight weight in kilograms will be collected to calculate body mass index. Weight and height will be combined to report BMI in kg/m^2.
Height | from enrollment at 12 month
  Height in meters will be collected to calculate body mass index. Weight and height will be combined to report BMI in kg/m^2.
Total cholesterol level | from enrollment at 12 month
  Total cholesterol level will be collected to check lipid levels
Total triglyceride level | from enrollment at 12 month
  Total triglyceride level will be collected to check lipid levels.
Low-density lipoprotein level | from enrollment at 12 month
  Low-density lipoprotein level will be collected to check lipid levels
High-density lipoprotein level | from enrollment at 12 month
  High-density lipoprotein level will be collected to check lipid levels.
Hemoglobin A1C level | from enrollment at 12 month
  Hemoglobin A1C level will be collected to check blood glucose.
Fasting glucose level | from enrollment at 12 month
  Fasting glucose level will be collected to check blood glucose.
Visit to general outpatient clinics (GOPC) | from enrollment at 12-month
  Visits to GOPC will be retrieved from the computerised clinical management system (CMS). This is to measure healthcare utilization.
Visit to emergency department | from enrollment at 12-month
  Visit to emergency department will be retrieved from the computerised clinical management system (CMS). This is to measure healthcare utilization.
Hospitalization | from enrollment at 12-month
  Hospitalization will be retrieved from the computerised clinical management system (CMS). This is to measure healthcare utilization.
Visits to private hospitals | from enrollment at 12-month
  Visits to private hospitals will be self-reported. This is to measure healthcare utilization.
Visits to private clinics | from enrollment at 12-month
  Visits to private clinics will be self-reported. This is to measure healthcare utilization.
Number of antihypertensive drug use | from enrollment at 12-month
  Number of antihypertensive drug use will be retrieved from the computerised clinical management system. This is to measure healthcare utilization.
Type of antihypertensive drug use | from enrollment at 12-month
  Type of antihypertensive drug use will be retrieved from the computerised clinical management system. This is to measure healthcare utilization.
Patients' productivity loss | from enrollment at 12-month
  Patients' productivity loss (e.g. loss of work days due to doctors' visits) will be self-reported.

CONTACTS AND LOCATIONS:
Locations (1):
- HKW and NTEC GOPC, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
May be available after discussion with other researchers

REFERENCES:
- [Derived] Ng SN, Yip BH, Wang S, Leung M, Choi SYK, Leung SY, Han JJ, Tsui WW, Lai SY, Chan L, Mihailidou AS, McManus RJ, Sy J, Lee EK. Can TElemedicine system replace doctor consultations to Achieve non-inferior blood pressure in patients with Controlled Hypertension (TEACH)? Study protocol for a randomised controlled trial. Trials. 2025 Dec 8;27(1):31. doi: 10.1186/s13063-025-09350-3. PMID 41361824